CLINICAL TRIAL: NCT04118504
Title: Randomised Controlled Clinical Trial of Intervention in Lifestyle and Therapeutic Adherence After Coronary Event Based on Interactive Web Application
Brief Title: Intervention in Lifestyle and Therapeutic Adherence After Coronary Event Based on Web Application
Acronym: EVITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI-0067-2018
Record Dates: First submitted 2019-09-30; First posted 2019-10-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Coronary Disease
Keywords: Coronary disease; Life style; Mobile application; Clinical trial
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Lifestyle intervention on through mobile application
  Interventions: Device: Mobile application
- Control group (No Intervention): Usual care

INTERVENTIONS:
Device: Mobile application — Lifestyle intervention on through mobile application
  Arms: Intervention group

SUMMARY:
Ischemic heart disease is the most frequent cause of mortality in the surrounding countries. Once a coronary event is over, there is a high risk of readmission, recurrence and, mortality, attributed to a sub-optimal control of cardiovascular risk factors (CVRF), highlighting the need to improve secondary prevention strategies aimed at changing lifestyle and therapeutic adherence. Preventive measures should be initiated during hospitalization as recommended by the clinical guidelines. The objective of this study is to evaluate, through a randomized controlled clinical trial, the effect of an intervention based on a web application of health (e-Health) on lifestyle (diet, physical activity and tobacco consumption) and medication adherence in people with coronary heart disease after percutaneous coronary intervention.

The sample will consist of 240 participants, 120 in the intervention group and 120 in the usual care group that will be evaluated at the beginning and nine months after hospital discharge regarding sociodemographic, clinical, CVRF, lifestyle and therapeutic adherence characteristics. The educational intervention, monitoring and self-monitoring will be carried out using a web-based e-Health tool, mobile phone application. The quantitative primary results will be compared between the two groups using ANCOVA adjusting for age and sex. Multivariate analysis will be carried out to examine the association of the intervention with life habits, control of CVRF, as well as with the evolution after discharge in respect of cardiovascular events, emergency and re-entry views.

DETAILED DESCRIPTION:
Design

1. A randomized single-blind, parallel-group, controlled clinical trial performed on patients with coronary heart disease who underwent a percutaneous coronary intervention (PCI) with stent placement in the Cardiology Service of a public reference hospital complex providing specialist care in the province of Cadiz, Spain, in which 1500 coronary interventions procedures are performed per year.
2. Randomization and Blinding The randomization and allocation to each group (1:1, intervention and usual care) are based on computer-generated random numbers. The researchers responsible for the study do not participate in the allocation of the participants. Due to the kind of intervention, blinding is not possible when the participants are allocated to groups. To minimize any bias, objective clinical variables are measured in the evaluation visit and the analyses are performed by blinded researchers.
3. Study Sample The participants are eligible to participate if they have a confirmed diagnosis of coronary heart disease and undergo stenting with PCI. Furthermore, the participants must comply with the criteria explained in the section.
4. Sample Size To detect a medium effect size of Cohen's d of 0.5 regarding adherence to the Mediterranean diet (8.6 ± 2.0 puntos), food consumption, vegetables (471.4 g/day ± 230.0 g/day), fruit (308.4 g/day ± 188.6 g/day), meat and derived products (149.7 g/day ± 63.7 g/day), fish (122.3 g/day ± 73.5 g/day), physical activity (210.2 METs-min/day -metabolic equivalents- ±221.8 METs-min/day) and a 12% decrease in smoking habits (prevalence of 21% in pilot study), a 95% confidence interval and a power of 90%, the sample size is estimated at 100 patients in each group. Assuming a 20% loss to follow-up with 240 participants, 120 in each arm: intervention and usual care.
5. Recruitment After the PCI and during admission, the nurse will recruit eligible patients and their care partners, will ask them to sign the informed consent, perform the initial assessment and organize a programmed visit after 36 weeks. A card will be provided with the date of the appointment and a telephone number for any changes.

   The participants allocated to the usual care group receive the standard prescribed care and advice about medication, and lifestyle.

   Both groups will be provided with written recommendations and an explanation about the standard Mediterranean diet, physical activity, stopping smoking and treatment adherence.

   Before hospital discharge, all the patients will be encouraged to follow a healthy lifestyle. Stages of change strategies will be used in addition to a motivational and behavior changing interview. Written information will be provided about risk factors, lifestyle goals, a suggested healthy menu, recommendations about the daily intake of food groups, and the other behavior that the intervention is targeting.
6. Intervention The intervention begins during the patient's stay in hospital immediately after a coronary event. The participants from the intervention group and their partner/carer will complete a short online tutorial describing the mobile application accessed using a mobile telephone or tablet. They will be advised to use the application for at least 15 min per day. This time has been considered sufficient for the daily recording of data in the pilot study. The intervention will last 36 weeks. If the patient does not record data for a week, he/she receives a message through the app encouraging him to use it. The patients may resolve any queries using the application's built-in messaging function, to which the nurse will reply through this messaging service or with a telephone call. This avoids many patient visits to the doctor for consultations and reduces human resource needs.

   Before the trial, a pilot study was performed with 20 participants to test the application and make any necessary adjustments.
7. Technical Data of the Website and Application The responsive online application (user registration, data management, downloading records) is managed via the project website, which acts as an access platform after validation with a password. The web environment enables the application to be executed using any browser. Operating environment: it is an application with remote access to a MySQL (My Structured Query Language) database. Technology development: (a) uses PHP scripting language (Personal Home Page Tools); (b) Asynchronous JavaScript and XML (AJAX) web development techniques . The application runs in the user's browser while it communicates with the server in the background; and (c) Bootstrap open-source tools for designing websites and online applications. Data storage: MySQL database is fast enough to deploy web applications. Data protection: in addition to on-demand backups performed by the software, the web server performs daily backups of all the files, so the data and program are doubly protected. Access privacy: The data are not stored in a local computer but on a web server, meaning they can only be accessed with a password. This web server works with anonymous data and is located in the country to comply with the regulations for the protection of high-level data.
8. Application Contents The application allows users to set goals and monitor their food consumption, physical exercise, blood pressure, tobacco use, and compliance with their treatment. It is based on the phases of change theory (attention, retention, memory, action, and motivation) and on making the process pleasing. The user's attention is caught through warnings and bright, attractive colors on the user interface; retention is encouraged by reminders, repetition and graphs; action is prompted by instructions, advice, and feedback; and motivation to change is boosted by internal comparisons (progress graphs), setting goals, self-monitoring and feedback.

   Through its different components (website, messages, emails, and calls), participants are encouraged to (1) follow a healthy eating pattern based on the Mediterranean diet aligned with national dietary guidelines; (2) perform physical activity of duration and intensity in line with the recommendations of their cardiologist; (3) stop smoking; (4) monitor their blood pressure; (5) adhere to their treatment by associating taking medication with daily activities, establishing set times for taking it and with support from a relative, etc.
9. Components of the Application A. Provide information encouraging a healthy lifestyle. Through the website the participants will have access to information on their screens that they can print to help them plan a healthier lifestyle and adhere to their treatment. The application also has a training section for the patient with information about the recommended therapeutic objectives in the clinical practice guidelines regarding food, physical activity, body weight, blood pressure, blood sugar, stopping smoking and adhering to treatment.

   B. Self-monitoring. The application has a recording and self-checking function to help patients to self-monitor the skills for each behavioral goal about nutrition, physical activity, tobacco consumption, blood pressure, body weight, capillary blood glucose in patients with diabetes mellitus and treatment adherence.
10. Training Session about the Application for Patient and Carer The nurse will install the shortcut to the application on the screen of the participant's mobile phone and will record the prescribed treatment including the name, dose, and timetable in the application. The nurse will update the prescription in the application if the doctor changes the treatment. During the training session, the participants learn to use the functions of the application: confirm when medication is taken, record the food consumed and physical activity performed (daily), blood pressure, weight, and tobacco consumption (weekly), and capillary blood glucose in participants with diabetes mellitus (twice a week).

    The participants can follow their evolution and progress through the graphics generated with the information they have recorded over the previous eight weeks.
11. Ethical Considerations The study will be conducted in agreement with the guidelines and protocols established in the Helsinki Declaration as revised in Fortaleza (Brazil) in October 2013, and complies with Law 14/2007 on Biomedical Research and with European Data Protection Regulations. It was approved by the Biomedical Research Ethics Committee of the Costa del Sol, Andalusian, with the reference: 003_ene19_PI-EVITE-18. The informed written consent of all the patients will be requested. The application guarantees the security measures regarding the current General Data Protection Regulations in Europe. It also includes data encryption mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Participants with coronary heart disease
* Under the age of 75
* Have a mobile phone

  * with the ability to receive text messages
  * with internet access

Exclusion Criteria:

* Severe heart failure
* Physical disability
* Dementia
* Congenital heart disease
* Rheumatic etiology disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet | 9 months
  14-item Questionnaire of Mediterranean diet adherence (unit of measure: points. Each item is scored 0 or 1. The total Mediterranean diet score ranges from 0 to 14 points. The higher the score, the higher the degree of adherence to the Mediterranean Diet.
Frequency of food consumption | 9 months
  Food-frequency questionnaire with 137 food items (unit of measure: number of times per month, week and day)
Level of physical activity | 9 months
  Minnesota Leisure Time Physical Activity Questionnaire (unit of measure: Metabolic equivalents-minutes per day. Minimum: 150 metabolic equivalents-minutes per day; active, those with energy expenditure in physical activity equal or greater than 150 metabolic equivalents-minutes per day). Do higher values represent a better outcome.
The concentration of carbon monoxide in exhaled air | 9 months
  Smoking cessation: Value < 6 parts per million of carbon monoxide in exhaled air. Smoker: Value > 6 parts per million of carbon monoxide in exhaled air.
Therapeutic adherence | 9 months
  A 4 items questionnaire (Total score: 4 points. Good therapeutic adherence= 4 points.Poor therapeutic adherence= 1-3 points)
Knowledge about cardiovascular disease using a questionnaire | 9 months
  24-item questionnaire (scale 0-5 each item. Do higher values represent a better outcome)
Usability and satisfaction with the application: 22 item questionnaire | 9 months
  22 item questionnaire to assess user acceptability of mobile health interventions. (6-point scale, level of disagreement to agreement with each item concerning the usability of the apps. Do higher values represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: MJ Santi, MD, Principal Investigator — Instituto de investigación e innovación biomédica de Cádiz
Locations (1):
- Hospital Puerta del Mar, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernal-Jimenez MA, Calle G, Gutierrez Barrios A, Gheorghe LL, Cruz-Cobo C, Trujillo-Garrido N, Rodriguez-Martin A, Tur JA, Vazquez-Garcia R, Santi-Cano MJ. Effectiveness of an Interactive mHealth App (EVITE) in Improving Lifestyle After a Coronary Event: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Apr 22;12:e48756. doi: 10.2196/48756. PMID 38648103